CLINICAL TRIAL: NCT04332458
Title: Motivators and Barriers for Physical Activity in Patients With Minor Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Christina Kruuse, Professor, Herlev Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-20014119
Record Dates: First submitted 2020-03-30; First posted 2020-04-02 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Stroke, Ischemic
Keywords: physical activity; motivators for physical activity; barriers for physical activity; secondary stroke prevention
MeSH Terms: conditions — Ischemic Stroke; Motor Activity

STUDY DESIGN:
Intervention Model Description: Focus group interviewing a cohort of patients with stroke (one group with previous exercise experience and a group without)
Masking Description: none of the participants are blinded in the focus group interview
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with stroke without exercise experience (Other): Patients who are discharged from the hospital within one month after a minor stroke or TIA and are not offered physical rehabilitation afterwards
  Interventions: Behavioral: A focus group interview
- Patients with stroke with exercise experience (Other): Patients with a minor stroke who have participated in an exercise study (HITPALS)
  Interventions: Behavioral: A focus group interview

INTERVENTIONS:
Behavioral: A focus group interview — this is a qualitative study using focus group interviewing.

SUMMARY:
The aim of this study is to investigate motivators and barriers for physical activity in patients discharged from hospital for a minor stroke or TIA. The study has a qualitative research design and will be conducted by focus group interviews.

DETAILED DESCRIPTION:
Little is known about motivators and barriers for physical activity after hospital discharge for patients with a minor stroke or TIA. These patients have few and temporary symptoms and are therefore discharged early from the hospital or seen in a outpatient TIA clinic. Standard treatment are preventive medication and advice on self-managed lifestyle changes. Occurrence of one ischemic stroke or TIA predisposes to further ischemic strokes and patients are at risk of developing cognitive deficits or vascular dementia over time unless multiple preventive measures are taken including physical activity. The purpose is to investigate motivators and barriers for physical activity after hospital discharge by focus-group interviewing this potential fragile group of patients. The research team want to facilitate the patients to be physically active and thereby prevent a recurrent stroke and slow the progression of vascular diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ischemic stroke or transient ischemic attack (TIA) without the need of a re-habilitation plan, but needs an exercise plan in order to prevent a recurrent stroke
* Patients who have participated in ≤ 1 hour of vigorous intensity activity on weekly basis within the last 3 months
* Patients able to speak, read, and understand Danish
* Patients ≥ 18 years of age and able to give informed consent

Exclusion Criteria:

* Patients with previous large artery stroke with sequelae preventing aerobic exercise in groups
* Symptoms or comorbidities preventing aerobic exercise in groups
* Dyspnoea caused by heart or lung diseases (e.g. chronic obstructive pulmonary disease (COPD))
* Aphasia or dementia interfering with participation in aerobic groups exercise
* Patients with Intermittent claudication/vascular claudication

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-03-21 (Actual); Study Completion 2022-01-16 (Actual)

PRIMARY OUTCOMES:
Motivators for physical activity | through study completion, an average of 1 year
  The study has a qualitative research design using focus group interviewing
Barriers for physical activity | through study completion, an average of 1 year
  The study has a qualitative research design using focus group interviewing

CONTACTS AND LOCATIONS:
Overall Officials: christina Kruuse, Professor, Principal Investigator — Herlev Gentofte Hospital, Department of Neurology
Locations (1):
- Herlev Hospital, Copenhagen, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No
Individual participant´s data cannot be shared with 3rd parties as these data are protected by Danish law